CLINICAL TRIAL: NCT06376578
Title: Comparing a Technology-enabled, Remotely Delivered Exercise Intervention to Partly-supervised Structured Exercise in Breast Cancer Survivors: a Randomised and Controlled Non- Inferiority Trial
Brief Title: Exercise Interventions for Improving Health in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Turner, Ph.D., FHEA, Dr James Turner, University of Bath
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 245256
Record Dates: First submitted 2020-11-20; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partly supervised, prescribed exercise group (Experimental): The partly-supervised, prescribed exercise group will be required to undertake two supervised exercise sessions and one unsupervised exercise session at home or in your local area each week. Supervised sessions will consist of exercising on both a treadmill and a stationary exercise bike. The intervention will be progressive, increasing in intensity and duration.
  Interventions: Behavioral: Exercise intervention
- Technology enabled, remotely delivered exercise group (Experimental): The technology enabled, remotely delivered exercise group will receive information and advice about exercise that could be undertaken at home or in their local area. In addition, participants will received a Polar A370 fitness tracker wristwatch with heart rate monitoring chest strap. Participants will take part in exercise each week (most likely walking) which will increase in duration over 8-weeks from 105 minutes each week to 150 minutes each week. Each week a member of the research team will have a telephone call with the participant to discuss the exercise prescription.
  Interventions: Behavioral: Polar A380 wristwatch physical activity tracker

INTERVENTIONS:
Behavioral: Exercise intervention — Exercise training will progress incrementally, increasing the duration of exercise on the treadmill by 5 minutes every 2 weeks whereby the final duration on the treadmill will be 35 minutes and the total duration will map onto recommended guidelines of 150 minutes per week. Throughout the 8-weeks, the duration of exercise on the cycle ergometer will remain at 15 minutes. Exercise intensity will progress throughout the 8-week intervention on both the treadmill and the cycle ergometer by 5% every 2 weeks, whereby exercise during the final week will be at 70% VO2max.
  Arms: Partly supervised, prescribed exercise group
Behavioral: Polar A380 wristwatch physical activity tracker — The research team will monitor individual exercise training weekly using virtual/electronic methods and a 30 minute telephone call. The researcher will provide feedback about how the participant's activity compares to physical activity recommendations, and encouragement and support will be provided verbally.
  Arms: Technology enabled, remotely delivered exercise group

SUMMARY:
Supervised, prescribed exercise has positive effects on body composition, physical functioning, psychological wellbeing and quality of life for patients after breast cancer treatment. However, exercise interventions are often time consuming, commonly take place at a health or fitness facility, and usually require a trained professional to be present. Cost-effective, enjoyable and practical approaches, that can be adopted at home or in local surroundings are needed. For example, an alternative approach is using an electronic physical activity tracking wristwatch to help patients engage with exercise or physical activity. Research demonstrates the importance of structured and supervised exercise for breast cancer survivors. However, it is not known whether other approaches (e.g. home-based exercise and physical activity) alongside the use of personalised technology-enabled feedback, can cause similar improvements to health when compared to structured exercise. The overall aim of this study is to determine whether cardiorespiratory fitness is changed by a technology enabled, remotely delivered exercise intervention and to determine whether this change is similar to the change caused by a partly supervised, prescribed exercise intervention. This study will also determine the influence of both interventions on physical functioning, body composition and blood pressure.

DETAILED DESCRIPTION:
Intervention groups:

Remotely-supported exercise group:

The remotely-supported group will received a target for a total duration of exercise each week (outdoor walking) progressing in duration from 105 to 150-min and 55% to 70% of V̇O2max. By week 7, the exercise prescription will align with common physical activity recommendations. Participants will be advised how they can break down their target into manageable bouts (e.g., 3 × 35 min walks = 105-min in week 1) and will be instructed to accumulate exercise with a minimum bout-length of 10-min. Intensity will be checked by participants using heart-rate thresholds that corresponded to their V̇O2max. Participants will take part in a weekly 30-min telephone calls to discuss the exercise they have completed, as documented by an internet-based data visualisation platform with data input from a wrist worn fitness tracker that records accelerometry data and heart rate

Partly-supervised exercise group:

The partly-supervised exercise group will undertake 2 supervised (laboratory-based treadmill and cycle ergometer exercise) and 1 unsupervised session per week (e.g., outdoor walking) progressing from 35 to 50-min and 55% to 70% of V̇O2max. By week 7, the exercise prescription will align with common physical activity recommendations. During supervised laboratory sessions, intensity will be confirmed and adjusted using indirect calorimetry. The intensity of unsupervised exercise sessions will be recorded using a chest-worn heart rate monitor.

Participant characterisation:

Participants will attend a laboratory for characterisation before and after the intervention (within 7 days) following a 10 hour overnight fast and after refraining from exercise, alcohol, and caffeine in the prior 24 hours. Body mass and height will be measured with the participant wearing light clothing. Body composition monitor. Dual-energy X-ray absorptiometry will be used to quantify fat mass, lean mass, and bone mineral density parameters. Blood pressure will be measured using an automated sphygmomanometer following 15 minutes rest in the supine position.

Physical function will be assessed using three tests. First, the 6-minute walk test, whereby participants will walk as far as possible in 6-minutes between two cones placed 7 meters apart. Second, the sit to stand test, whereby participants will perform as many sit-to-stands as possible in 30 seconds (i.e., seated on a standardised chair, rising to reach full knee extension, returning to a seated position, arms folded across the chest). Third, the 8 foot up timed up and go test, whereby participants will rise from being in a seated position on a standardised chair, walk 8 feet, and return to a seated position as quickly as possible.

Cardiorespiratory fitness will be assessed using a treadmill-based maximal walking exercise test to exhaustion comprising 3-minute stages, beginning at 2.7 kph with a 1% gradient and increasing by 1.3 kph until 6.6 kph, with further intensity increments via increasing gradient by 2%. During the final minute of each stage, heart rate will be measured using telemetry and rating of perceived exertion will be recorded. Expired air samples will be collected using Douglas bags during the final minute of each stage. Oxygen and carbon dioxide within each bag will be analysed using a gas analyser and volume and temperature of the air will be assessed using a digital thermometer and dry gas meter.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-69 years
* History of previous stage I-III invasive breast cancer
* No history of metastatic cancer
* No significant cardiac co-morbidity
* No diagnosis of bilateral breast cancer
* > 2 months from surgery, chemotherapy and radiotherapy treatments, however patients continuing with endocrine therapy will be included.
* BMI 20 > <35 kg.m2
* Oncologist clearance
* Pass physical activity readiness questionnaire (PAR-Q)
* Last menstrual period >1 year ago

Exclusion Criteria:

* Current malignancy
* Previous superficial basal cell carcinoma of the skin or prior carcinoma-in situ (including ductal carcinoma in situ/lobular carcinoma in situ of breast) is allowed
* Cardiovascular Disease
* Severe hypertension (>200/120 mmHg)
* 5+ years since last treatment
* Active infection at recruitment
* Undertaking regular, structured, exercise training defined as self-reported structured physical activity lasting > 30 minutes on two or more occasions per week (measured before the first visit using the international physical activity questionnaire (IPAQ))
* Contraindication to undertaking an exercise programme including previously diagnosed significant osteoporosis or other co-morbidities at the oncologist's discretion

Ages: 35 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in VO2max (maximum oxygen uptake) | 9 weeks
  Measure of cardiorespiratory fitness

SECONDARY OUTCOMES:
Change in Body composition | 9 weeks
  Measured by Body Mass Index and Dual energy x-ray absorptiometry

OTHER OUTCOMES:
Change in physical functioning | 9 weeks
  Assessed by 6 minute walk test, 8 foot get up and go test, sit to stand test
Change in Psychological measures | 9 weeks
  Enjoyment, depression, anxiety and stress
Change in immune profiles and function | 9 weeks
  Leukocyte differential, lymphocyte phenotypes and function in blood

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Struszczak L, Walhin JP, Betts J, Thompson D, Beresford M, Turner JE. Cardiorespiratory Fitness, Functional Fitness and Body Composition Among Breast Cancer Survivors With 8 Weeks of Exercise Training: A Randomised, Controlled Non-Inferiority Trial Comparing Remotely-Supported and Partly-Supervised Interventions. Cancer Med. 2026 Feb;15(2):e71608. doi: 10.1002/cam4.71608. PMID 41656158